CLINICAL TRIAL: NCT03082729
Title: A Phase IV, Open Label Study of the Effects of Apremilast on Vascular Inflammation and Cardiometabolic Function in Psoriasis
Brief Title: Vascular Inflammation in Psoriasis - Apremilast
Acronym: VIP-A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Celgene Corporation (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 826652; 97509210 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2017-02-22; First posted 2017-03-17 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Psoriasis; Cardiovascular Diseases
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases | interventions — apremilast

STUDY DESIGN:
Masking Description: Imaging data files will be sent to the central core of the National Institutes of Health (NIH) Imaging Lab for measuring the standardized uptake values (SUVs). The NIH central PET/CT readers will be blinded to time point of scan via Digital Imaging and Communication in Medicine (DICOM) file editing applied by the University of Pennsylvania.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apremilast (Other): Apremilast (Otezla), 30mg oral tablet twice per day for 52 weeks. Single arm, open label study.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast (brand name Otezla) is a medication for the treatment of certain types of psoriasis and psoriatic arthritis.
  Other Names: Otezla

SUMMARY:
The purpose of the VIP-A study is to determine the effect of apremilast on aortic vascular inflammation, cardiometabolic biomarkers and body composition in patients with moderate-severe psoriasis.

DETAILED DESCRIPTION:
The primary objectives of this study are to determine the effect of apremilast on aortic vascular inflammation, cardiometabolic biomarkers and body composition in patients with moderate-severe psoriasis. Fluorodeoxyglucose (FDG) - positron emission tomography (PET)/computed tomography (CT) will be used to assess vascular inflammation, with multi-volumetric product, tissue-to-background ratio and total atherosclerotic burden, and body composition via volumetric quantification. This is a year-long, single arm, open label study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age and older.
* Clinical diagnosis of psoriasis for at least 6 months as determined by medical history interview and confirmation of diagnosis through physical examination by Investigator.
* Stable plaque psoriasis for at least 2 months before screening and at baseline (Week 0) as determined by medical history interview.
* Moderate to severe psoriasis defined by ≥ 10 percent Body Surface Area (BSA) involvement at the baseline (Week 0) visit.
* Psoriasis Area and Severity Index (PASI) score of ≥ 12 at the Baseline (Week 0) visit.
* Participant is a candidate for systemic therapy and has active psoriasis despite prior treatment with topical agents.
* Women are eligible to participate in the study if they meet one of the following criteria:
* Females of childbearing potential (FCBP) must have a negative pregnancy test at screening and baseline. Women of childbearing potential must undergo periodic pregnancy testing during the study and agree to use at least one of the following methods of contraception throughout the study duration and for at least 28 days after taking the last dose of investigational product:
* Oral contraceptives
* Transdermal contraceptives
* Injectable or implantable methods
* Intrauterine devices
* Vaginal ring
* Vasectomized partner
* Barrier methods (Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.);
* Women who are postmenopausal (for at least one year), sterile, or hysterectomized;
* Women who have undergone tubal ligation will be required to undergo periodic pregnancy testing during the duration of the study
* Sexual abstinence, defined as total abstinence from sexual intercourse, is considered an adequate form of contraception. (Agreement to comply with sexual abstinence must be recorded in the source document).
* Participants using oral or parenteral forms of contraceptives must have been using these methods for at least 90 days prior to baseline visit.
* Men (including those who have had a vasectomy), who engage in activity in which conception is possible, are eligible to participate if they:
* Use barrier contraception (male latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.
* Participant is judged to be in good general health as determined by the Principal Investigator based upon the results of medical history, laboratory profile and physical examination performed at screening.

Exclusion Criteria:

* Prior treatment with apremilast.
* Diagnosis of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.
* Diagnosis of other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis.
* Cannot avoid topical prescription medications for psoriasis for at least 14 days prior to the baseline visit (week 0) and during the study, with the exception of hydrocortisone 2.5% for the face and intertriginous areas.
* Cannot avoid ultraviolet B (UVB) phototherapy or Excimer laser for at least 14 days prior to the Baseline (Week 0) visit and during the study.
* Cannot avoid psoralen-ultraviolet A (UVA) phototherapy for at least 30 days prior to the Baseline (Week 0) visit and during the study.
* Use of systemic therapies for the treatment of psoriasis, or systemic therapies known to improve psoriasis, during the study:
* Systemic therapies must be discontinued at least 30 days prior to the Baseline (Week 0) visit except for biologics.
* All biologics, except interleukin (IL)-12/IL-23 antagonists, must be discontinued for at least 90 days prior to Baseline (Week 0).
* Any IL-12/IL-23 antagonist (e.g., ustekinumab, briakinumab) must be discontinued for at least 180 days prior to Baseline (Week 0).
* Investigational agents must be discontinued at least 30 days or 5 half-lives (whichever is longer) prior to the Baseline (Week 0) visit.
* Participant is ≥ 300lbs
* Participant is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.
* Participant is taking a medication that interferes with metabolism of apremilast, including but not limited to rifampin, phenobarbital, carbamazepine, phenytoin
* Poorly controlled medical condition, such as unstable ischemic heart disease, cerebrovascular accident or myocardial infarction within the prior 6 months, psychiatric disease requiring frequent hospitalization, and any other condition, which, in the opinion of the Investigator, would put the participant at risk by participation in the study.
* Prior history of suicide attempt at any time in the participant's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Uncontrolled hypertension, with measured systolic blood pressure >180 mmHg or diastolic blood pressure >95 mmHg
* Participant has infection or risk factors for severe infections, for example
* Positive serology or known history of HIV, hepatitis B or C, or other severe, recurrent, or persistent infections;
* Excessive immunosuppression or other factors associated with it, including human immunodeficiency virus infection;
* Active tuberculosis (TB) disease;
* Any other significant infection requiring hospitalization or intravenous (IV) antibiotics in the 30 days prior to baseline;
* Infection requiring treatment with oral or parenteral (other than IV) antibiotics within 14 days prior to baseline;
* Participant has received vaccination with a live viral agent within 30 days prior to screening or will require a live vaccination during study participation including up to 30 days after the last dose of study drug.
* Participant has history of hematological or solid malignancy other than successfully treated basal cell carcinoma, non-metastatic cutaneous squamous cell carcinoma or cervical intraepithelial neoplasia or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
* Female participant who is pregnant or breast-feeding or considering becoming pregnant during the study.
* Screening clinical laboratory analyses showing any of the following abnormal results:
* White blood cell (WBC) count <3.0 x 109/L. (Subject can be included if WBC count is <3.0 x 109/L and absolute neutrophil count (ANC) is >1000 cells / mm3.)
* WBC count > 15 x 109/L;
* Hemoglobin (Hgb) < 9.0 x 109/L;
* Platelet count < 100 x 109/L;
* Serum creatinine >1.5 mg/dL ;
* Serum aspartate transaminase or alanine transaminase >2.0 upper limits of normal
* Recent history of substance abuse or psychiatric illness that could preclude compliance with the protocol.
* History of substance abuse within 365 days of screening visit.
* Alcohol use of more than 14 drinks per week within 14 days of the baseline visit
* If subject is on cholesterol-lowering medication (e.g. statin), dose and form of medication must be stable for 90 days prior to week 0 and remain stable throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males and females 18 years of age and older.
Enrollment: 70 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Southern California, Los Angeles, California
  - Derm Associates, P.C., Rockville, Maryland
  - Buffalo Medical Group, P.C., Buffalo, New York
  - Oregon Medical Research Center, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Center for Clinical Studies, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gelfand JM, Shin DB, Armstrong AW, Tyring SK, Blauvelt A, Gottlieb S, Lockshin BN, Kalb RE, Fitzsimmons R, Rodante J, Parel P, Manyak GA, Mendelsohn L, Noe MH, Papadopoulos M, Syed MN, Werner TJ, Wan J, Playford MP, Alavi A, Mehta NN. Association of Apremilast With Vascular Inflammation and Cardiometabolic Function in Patients With Psoriasis: The VIP-A Phase 4, Open-label, Nonrandomized Clinical Trial. JAMA Dermatol. 2022 Dec 1;158(12):1394-1403. doi: 10.1001/jamadermatol.2022.3862. PMID 36129688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and one patients were screened, and 70 patients met inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Apremilast
Started | 70
Per Protocol Population Week 16 | 60
Completed | 39
Not Completed | 31
Not completed — Lost to Follow-up | 7
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 9
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 6
Not completed — Fear of study procedure | 1
Not completed — Scheduling conflict | 1

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.47 (14.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 58
  More than one race | 4
  Unknown or Not Reported | 0
Drink alcohol [Count of Participants; unit: Participants]
  Yes | 39
  No | 31
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 17
  Former smoker | 23
  Never smoked | 30
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.22 (5.02)
Weight [Mean (Standard Deviation); unit: kg] | 90.36 (17.41)
Medical history [Count of Participants; unit: Participants]
  Diabetes | 6
  Hyperlipidemia | 16
  Hypertension | 19
  Statin use | 12
Age at psoriasis diagnosis [Mean (Standard Deviation); unit: years] | 31.21 (16.86)
History of psoriatic arthritis [Count of Participants; unit: Participants] | 8
Psoriasis treatment history [Count of Participants; unit: Participants]
  Any phototherapy | 21
  Any oral systemics | 24
  Any biologics | 30
  Any investigational agents | 7
Baseline PASI [Mean (Standard Deviation); unit: units on a scale] — Psoriasis Area and Severity Index (PASI) is the most widely used tool for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
  units on a scale | 18.62 (5.96)
Baseline PGA [Mean (Standard Deviation); unit: score on a scale] — Physician Global Assessment (PGA) is calculated by averaging three subcomponent scores (induration, erythema, and scaling) that are graded from 0 (no involvement) to 5 (maximum involvement) that are averaged over all psoriatic lesions.
  score on a scale | 0.32 (0.54)
Baseline DLQI [Mean (Standard Deviation); unit: score on a scale] — The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. The score ranges from 0 to 30; 0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect.
  score on a scale | 11.60 (6.72)
Baseline Pruritus VAS [Mean (Standard Deviation); unit: units on a scale] — A visual analogue scale for pruritus (itch), ranging from 0 (no itch) to 100 (worst imaginable itch).
  units on a scale | 57.18 (30.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Vascular Inflammation of the Aorta as Measured by FDG-PET/CT Between Baseline and Week 16.
Description: The primary analysis will consist of comparisons of total vascular inflammation of the aorta between week 16 and baseline using [18F]-Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) / Computed Tomography (CT) (FDG-PET/CT). Tissue-to-background ratio (TBR) of the standardized uptake value (SUV) is used to assess the level of inflammation of the aorta relative to the venous blood pool (background reference).
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Apremilast
Number analyzed (Participants) | 57
ratio | -0.017 (0.033)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.612, t-test, 2 sided

2. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Ferritin
Description: Ferritin is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
ng/ml | -13.416 (7.614)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.083, t-test, 2 sided

3. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: C Reactive Protein (CRP)
Description: CRP is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µg/ml | -414.175 (823.144)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.617, t-test, 2 sided

4. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Intercellular Adhesion Molecule (ICAM)-1
Description: ICAM-1 is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µg/ml | -169.902 (264.980)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.524, t-test, 2 sided

5. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Serum Amyloid-A (SAA)
Description: SAA is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µg/ml | 46.047 (1324.285)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.972, t-test, 2 sided

6. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Vascular Cell Adhesion Molecule (VCAM)-1
Description: VCAM-1 is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µg/ml | -11.201 (11.061)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.315, t-test, 2 sided

7. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Interferon (IFN)-Gamma
Description: IFN-gamma is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | -1.944 (2.514)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.443, t-test, 2 sided

8. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Interleukin (IL)-1b
Description: IL-1b is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | -0.472 (0.208)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.027, t-test, 2 sided

9. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: IL-10
Description: IL-10 is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | -0.054 (0.063)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.390, t-test, 2 sided

10. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: IL-17A
Description: IL-17A is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | -0.947 (0.593)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.116, t-test, 2 sided

11. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: IL-6
Description: IL-6 is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | 2.727 (2.779)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.331, t-test, 2 sided

12. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: IL-8
Description: IL-8 is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | 24.014 (19.571)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.225, t-test, 2 sided

13. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: IL-9
Description: IL-9 is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | -0.090 (0.061)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.141, t-test, 2 sided

14. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Monocyte Chemoattractant Protein (MCP)-1
Description: MCP-1 is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | 3.056 (20.557)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.882, t-test, 2 sided

15. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Tumor Necrosis Factor (TNF)-Alpha
Description: TNF-alpha is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
pg/ml | 17.914 (18.095)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.326, t-test, 2 sided

16. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: IL2RA
Description: IL2RA is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
ng/ml | -3.308 (1.940)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.094, t-test, 2 sided

17. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: GlycA
Description: GlycA is a marker of inflammation.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | 10.690 (6.145)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.087, t-test, 2 sided

18. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Cholesterol Efflux Capacity
Description: Cholesterol Efflux Capacity is a marker of lipid function and metabolism.
  The ability to promote cholesterol efflux from macrophages is a classic function of HDL that is thought to be an important mechanism by which HDL protects against atherosclerosis. HDL cholesterol efflux capacity assays are performed based on published methods using J774 cells derived from a murine macrophage cell line (Mehta NN Atherosclerosis 2012). Efflux is calculated as a unitless measure by using the following formula: [(µCi of 3H-cholesterol in media containing apoB-depleted subject plasma - µCi of 3H-cholesterol in plasma-free media) / (µCi of 3H-cholesterol in media containing apoB-depleted pooled control plasma-µCi of 3H-cholesterol in pooled control plasma-free media)]. Cholesterol efflux capacity is inversely correlated with incidence of cardiovascular events (i.e. higher cholesterol efflux capacity is better for patients).
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: unitless measure
Arm/Group | Apremilast
Number analyzed (Participants) | 59
unitless measure | -0.010 (0.033)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.771, t-test, 2 sided

19. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Triglyceride
Description: Triglyceride is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 59
mg/dL | -3.542 (5.108)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.491, t-test, 2 sided

20. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Total Cholesterol
Description: Total Cholesterol is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 59
mg/dL | 0.254 (2.663)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.924, t-test, 2 sided

21. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: High-density Lipoprotein (HDL) - Cholesterol (C)
Description: HDL-C is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 59
mg/dL | 0.136 (0.812)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.868, t-test, 2 sided

22. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: HDL-Particle Number (P)
Description: HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µmol/L | 0.058 (0.585)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.922, t-test, 2 sided

23. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: HDL-Particle Size (Z)
Description: HDL-Z is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Measure: Mean (Standard Error); unit: nm
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nm | -0.071 (0.054)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.192, t-test, 2 sided

24. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Small (S)-HDL-P
Description: S-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µmol/L | 0.507 (0.671)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.453, t-test, 2 sided

25. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Medium (M)-HDL-P
Description: M-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µmol/L | -0.203 (0.553)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.714, t-test, 2 sided

26. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Large and Medium (LM)-HDL-P
Description: LM-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µmol/L | -0.442 (0.561)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.434, t-test, 2 sided

27. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Large (L)-HDL-P
Description: L-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µmol/L | -0.231 (0.234)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.329, t-test, 2 sided

28. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Low-density Lipoprotein (LDL)-C
Description: LDL-C is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 59
mg/dL | 0.119 (2.549)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.963, t-test, 2 sided

29. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: LDL-P
Description: LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | -21.712 (25.618)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.400, t-test, 2 sided

30. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: LDL-Z
Description: LDL-Z is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nm
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nm | 0.086 (0.070)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.223, t-test, 2 sided

31. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: S-LDL-P
Description: S-LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | -31.780 (26.849)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.241, t-test, 2 sided

32. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: L-LDL-P
Description: L-LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µmol/L | 21.763 (23.001)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.348, t-test, 2 sided

33. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Very Large (VL)-LDL-P
Description: VL-LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | -18.678 (23.175)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.424, t-test, 2 sided

34. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Very Low-density Lipoprotein (VLDL)-P
Description: VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | 1.227 (2.842)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.667, t-test, 2 sided

35. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: VLDL-Z
Description: VLDL-Z is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nm
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nm | -1.607 (1.060)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.135, t-test, 2 sided

36. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: VLDL-Triglycerides (TG)
Description: VLDL-TG is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 59
mg/dL | -4.393 (4.480)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.331, t-test, 2 sided

37. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: S-VLDL-P
Description: S-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | 1.371 (2.212)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.538, t-test, 2 sided

38. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: M-VLDL-P
Description: M-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | 0.625 (2.351)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.791, t-test, 2 sided

39. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: LM-VLDL-P
Description: LM-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | -0.214 (2.245)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.925, t-test, 2 sided

40. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: L-VLDL-P
Description: L-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | -0.900 (0.633)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.161, t-test, 2 sided

41. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Intermediate-density Lipoprotein (IDL)-P
Description: IDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 59
nmol/L | -11.763 (19.357)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.546, t-test, 2 sided

42. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Apolipoprotein A1 (ApoA1)
Description: ApoA1 is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 58
mg/dL | 0.939 (2.170)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.667, t-test, 2 sided

43. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Apolipoprotein B (ApoB)
Description: ApoB is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 58
mg/dL | 0.308 (1.519)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.840, t-test, 2 sided

44. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: TRLTG
Description: TRLTG is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 58
mg/dL | -5.142 (5.655)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.367, t-test, 2 sided

45. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: (Triglyceride-Rich Lipoprotein Cholesterol) TRLC
Description: TRLC is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 58
mg/dL | -0.352 (1.215)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.773, t-test, 2 sided

46. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: (Triglyceride-Rich Lipoprotein) TRLP
Description: TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
nmol/L | 0.283 (6.945)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.968, t-test, 2 sided

47. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: VS-TRLP
Description: VS-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
nmol/L | 0.445 (7.569)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.953, t-test, 2 sided

48. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: S-TRLP
Description: S-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
nmol/L | 0.534 (4.778)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.911, t-test, 2 sided

49. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: M-TRLP
Description: M-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
nmol/L | 0.115 (1.616)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.944, t-test, 2 sided

50. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: L-TRLP
Description: L-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
nmol/L | -0.811 (0.663)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.226, t-test, 2 sided

51. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: VL-TRLP
Description: VL-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
nmol/L | -0.000 (0.009)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.988, t-test, 2 sided

52. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Insulin
Description: Insulin is a marker of glucose metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
ng/ml | 159.448 (120.095)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.189, t-test, 2 sided

53. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR is a marker of glucose metabolism. HOMA-IR, a method used to quantify insulin resistance and beta-cell function, is expressed using fasting blood glucose and insulin levels. It is calculated using the formula (HOMA-IR = fasting glucose [mg/dl] * fasting insulin [mU/ml]/405).
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: index
Arm/Group | Apremilast
Number analyzed (Participants) | 58
index | 0.551 (0.791)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.488, t-test, 2 sided

54. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Glucose
Description: Glucose is a marker of metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Apremilast
Number analyzed (Participants) | 58
mg/dL | 2.615 (4.074)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.523, t-test, 2 sided

55. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Diabetes Risk Index (DRI)
Description: DRI is a marker of glucose metabolism. DRI is a nuclear magnetic resonance spectroscopy (NMR)-derived multimarker score (values 1-100) that predicts a patient's risk of developing type 2 diabetes mellitus (T2D) independent of glycemic status. DRI derives its performance from the weighted addition of the Lipoprotein Insulin Resistance Index (LP-IR) scores with simultaneously-measured levels of branched-chain amino acids (BCAA). Higher scores indicate greater risk.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: index
Arm/Group | Apremilast
Number analyzed (Participants) | 58
index | -2.978 (1.551)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.060, t-test, 2 sided

56. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Lipoprotein Insulin Resistance Index (LP-IR)
Description: LP-IR is a marker of glucose metabolism. LP-IR is a marker of insulin resistance, and as such the LP-IR score predicts a patient's likelihood of future development of type 2 diabetes. LP-IR is a multimarker index (values 0-100) based on the concentrations of particular lipoprotein subclasses. Greater score indicates higher likelihood of developing diabetes.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: index
Arm/Group | Apremilast
Number analyzed (Participants) | 59
index | -0.763 (2.679)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.777, t-test, 2 sided

57. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Leptin
Description: Leptin is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
ng/ml | -84.193 (1232.360)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.946, t-test, 2 sided

58. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Adiponectin
Description: Adiponectin is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 59
µg/ml | -1.430 (1.521)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.351, t-test, 2 sided

59. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Fetuin A
Description: Fetuin A is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Apremilast
Number analyzed (Participants) | 57
µg/ml | -50.732 (24.231)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.041, t-test, 2 sided

60. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Citrate
Description: Citrate is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | 0.429 (2.921)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.884, t-test, 2 sided

61. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Valine
Description: Valine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -14.301 (5.858)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.018, t-test, 2 sided

62. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Leucine
Description: Leucine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -9.185 (4.509)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.046, t-test, 2 sided

63. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Isoleucine
Description: Isoleucine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -6.018 (2.462)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.018, t-test, 2 sided

64. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Alanine
Description: Alanine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -20.059 (18.497)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.283, t-test, 2 sided

65. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: BCAA
Description: Branched-chain amino acids (BCAA) is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -29.505 (11.118)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.010, t-test, 2 sided

66. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Ketone Bodies
Description: Ketone Bodies are markers of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -30.319 (33.598)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.371, t-test, 2 sided

67. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Beta Hydroxybutyrate
Description: Beta Hydroxybutyrate is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -13.859 (23.337)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.555, t-test, 2 sided

68. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Acetoacetic Acid
Description: Acetoacetic Acid is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | 0.711 (1.134)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.533, t-test, 2 sided

69. Primary Outcome: Changes in Cardiometabolic Markers Between Baseline and Week 16: Acetone
Description: Acetone is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 16 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Apremilast
Number analyzed (Participants) | 58
µmol/L | -17.171 (11.389)
Statistical Analysis 1: Comparison: Apremilast; Test type: Superiority; p = 0.137, t-test, 2 sided

70. Secondary Outcome: Changes in Body Composition as Measured by FDG-PET/CT Between Week 52 and and Earlier Time Points (Baseline and Week 16): Visceral Adipose Tissue
Description: Secondary analysis will consist of comparisons of change in body composition between weeks 52, 16, and baseline. Visceral adipose tissue quantification using a single CT slice at the level of the umbilicus using computer-assisted tissue segmentation (Pescatori LC et al. Quantification of visceral adipose tissue by computed tomography and magnetic resonance imaging: reproducibility and accuracy. Radiol Bras. 2019 15(1):1-6.).
  The values represent the cross-sectional area of the tissue segmented on the CT slice (cm^2); higher values indicate greater amount of visceral adipose tissue.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: cm^2
Groups:
- Week 16 vs. Baseline: Assessment of difference between Week 16 and Baseline
- Week 52 vs. Baseline: Assessment of difference between Week 52 and Baseline
- Week 52 vs. Week 16: Assessment of differences between Week 52 and Week 16
Arm/Group | Week 16 vs. Baseline | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 57 | 38 | 38
cm^2 | -10.681 (3.052) | -12.519 (4.898) | 2.189 (3.517)
Statistical Analysis 1: Comparison: Week 16 vs. Baseline; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.015, t-test, 2 sided
Statistical Analysis 3: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.537, t-test, 2 sided

71. Secondary Outcome: Changes in Body Composition as Measured by FDG-PET/CT Between Week 52 and and Earlier Time Points (Baseline and Week 16): Subcutaneous Adipose Tissue
Description: Secondary analysis will consist of comparisons of change in body composition between weeks 52, 16, and baseline. Subcutaneous adipose tissue quantification using a single CT slice at the level of the umbilicus using computer-assisted tissue segmentation (Pescatori LC et al. Quantification of visceral adipose tissue by computed tomography and magnetic resonance imaging: reproducibility and accuracy. Radiol Bras. 2019 15(1):1-6.).
  The values represent the cross-sectional area of the tissue segmented on the CT slice (cm^2); higher values indicate greater amount of subcutaneous adipose tissue.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | Week 16 vs. Baseline | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 57 | 38 | 38
cm^2 | -19.857 (5.405) | -19.585 (7.170) | 0.638 (6.133)
Statistical Analysis 1: Comparison: Week 16 vs. Baseline; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.010, t-test, 2 sided
Statistical Analysis 3: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.918, t-test, 2 sided

72. Secondary Outcome: Changes in Physician Reported Outcomes: Psoriasis Area and Severity Index (PASI)
Description: Secondary analysis will consist of comparisons of change in PASI scores. PASI is the most widely used tool for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Time Frame: Baseline, week 16, and week 52.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Week 52 vs. Baseline: Assessment of differences between Week 52 and Baseline
Arm/Group | Week 16 vs. Baseline | Week 52 vs. Baseline
Number analyzed (Participants) | 60 | 39
score on a scale | -10.778 (0.852) | -9.903 (1.095)
Statistical Analysis 1: Comparison: Week 16 vs. Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided

73. Secondary Outcome: Changes in Physician Reported Outcomes: Physician Global Assessment (PGA)
Description: Secondary analysis will consist of comparisons of change in PGA scores. Physician Global Assessment (PGA) is calculated by averaging three subcomponent scores (induration, erythema, and scaling) that are graded from 0 (no involvement) to 5 (maximum involvement) that are averaged over all psoriatic lesions. Higher scores indicate greater disease burden.
Time Frame: Baseline, week 16, and week 52.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Week 16 vs. Baseline | Week 52 vs. Baseline
Number analyzed (Participants) | 60 | 39
score on a scale | -1.200 (0.106) | -1.067 (0.169)
Statistical Analysis 1: Comparison: Week 16 vs. Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided

74. Secondary Outcome: Changes in Patient Reported Outcomes: Dermatology Life Quality Index (DLQI)
Description: Secondary analysis will consist of comparisons of change in DLQI scores. DLQI is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. The score ranges from 0 to 30; 0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect.
Time Frame: Baseline, week 16, and week 52.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Week 16 vs. Baseline | Week 52 vs. Baseline
Number analyzed (Participants) | 60 | 39
score on a scale | -6.050 (0.723) | -5.692 (1.125)
Statistical Analysis 1: Comparison: Week 16 vs. Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided

75. Secondary Outcome: Changes in Patient Reported Outcomes: Pruritis by Visual Analog Scales (VAS)
Description: Secondary analysis will consist of comparisons of change in Pruritus VAS scores.
  A visual analogue scale for pruritus (itch), ranging from 0 (no itch) to 100 (worst imaginable itch).
Time Frame: Baseline, week 16, and week 52.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Week 16 vs. Baseline | Week 52 vs. Baseline
Number analyzed (Participants) | 60 | 39
score on a scale | -27.527 (4.349) | -19.110 (6.249)
Statistical Analysis 1: Comparison: Week 16 vs. Baseline; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.004, t-test, 2 sided

76. Secondary Outcome: Change in Vascular Inflammation of the Five Aortic Segments as Measured by FDG-PET/CT Between Week 52, 16, and Baseline.
Description: Secondary analysis will consist of comparisons of vascular inflammation of the five aortic segments using TBR between week 52, 16, and baseline.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Week 16 vs. Baseline | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 57 | 38 | 38
ratio
  Ascending aorta | -0.067 (0.040) | -0.099 (0.046) | 0.028 (0.039)
  Aortic arch | -0.062 (0.036) | -0.080 (0.047) | 0.010 (0.036)
  Descending aorta | -0.000 (0.037) | -0.057 (0.041) | -0.019 (0.042)
  Abdominal aorta (suprarenal) | -0.026 (0.035) | -0.075 (0.042) | -0.017 (0.043)
  Abdominal aorta (infrarenal) | -0.030 (0.055) | -0.118 (0.073) | -0.038 (0.052)

77. Secondary Outcome: Change in Total Vascular Inflammation of the Aorta as Measured by FDG-PET/CT Between Week 52 and Earlier Time Points.
Description: Secondary analysis will consist of comparisons of total vascular inflammation of the aorta using TBR between week 52, 16, and baseline.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
ratio | -0.069 (0.040) | -0.016 (0.038)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.092, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.678, t-test, 2 sided

78. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Ferritin
Description: Ferritin is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
ng/ml | -22.645 (9.287) | -1.736 (5.680)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.020, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.762, t-test, 2 sided

79. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): CRP
Description: CRP is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µg/ml | 36.050 (1043.600) | -246.058 (988.627)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.973, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.805, t-test, 2 sided

80. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): ICAM-1
Description: ICAM-1 is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µg/ml | 41.059 (667.553) | 292.802 (662.249)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.951, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.661, t-test, 2 sided

81. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): SAA
Description: SAA is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µg/ml | 1586.025 (3114.549) | 2799.836 (2695.059)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.614, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.306, t-test, 2 sided

82. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): VCAM-1
Description: VCAM-1 is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µg/ml | 10.253 (10.220) | 24.967 (11.215)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.322, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.032, t-test, 2 sided

83. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IFN-gamma
Description: IFN-gamma is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | 0.281 (5.509) | 4.717 (4.194)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.960, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.268, t-test, 2 sided

84. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IL-1b
Description: IL-1b is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | 0.285 (0.419) | 0.624 (0.517)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.501, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.235, t-test, 2 sided

85. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IL-10
Description: IL-10 is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | 0.631 (0.551) | 0.689 (0.551)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.259, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.219, t-test, 2 sided

86. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IL-17A
Description: IL-17A is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | -1.383 (0.917) | 0.141 (0.294)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.140, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.633, t-test, 2 sided

87. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IL-6
Description: IL-6 is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | 22.680 (21.683) | 18.344 (21.769)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.302, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.405, t-test, 2 sided

88. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IL-8
Description: IL-8 is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | 369.437 (349.058) | 330.646 (330.466)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.297, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.324, t-test, 2 sided

89. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IL-9
Description: IL-9 is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | -0.025 (0.103) | 0.080 (0.070)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.812, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.264, t-test, 2 sided

90. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): MCP-1
Description: MCP-1 is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | 101.704 (93.377) | 78.605 (67.289)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.283, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.250, t-test, 2 sided

91. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): TNF-alpha
Description: TNF-alpha is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
pg/ml | 100.589 (71.944) | 72.650 (62.065)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.170, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.249, t-test, 2 sided

92. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IL2RA
Description: IL2RA is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
ng/ml | -1.557 (2.432) | 0.782 (1.618)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.526, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.632, t-test, 2 sided

93. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): GlycA
Description: GlycA is a marker of inflammation.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | 4.324 (7.836) | -8.703 (6.533)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.584, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.191, t-test, 2 sided

94. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Cholesterol Efflux Capacity
Description: as for outcome 18
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: unitless measure
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
unitless measure | -0.159 (0.053) | -0.111 (0.036)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.005, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.004, t-test, 2 sided

95. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Triglyceride
Description: Triglyceride is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
mg/dL | 4.684 (7.448) | 12.526 (6.936)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.533, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.079, t-test, 2 sided

96. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Total Cholesterol
Description: Total Cholesterol is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
mg/dL | 4.316 (4.447) | 7.474 (4.302)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.338, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.091, t-test, 2 sided

97. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): HDL-C
Description: HDL-C is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
mg/dL | 1.842 (1.100) | 1.711 (1.173)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.102, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.153, t-test, 2 sided

98. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): HDL-P
Description: HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µmol/L | 0.953 (0.774) | 1.092 (0.879)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.226, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.222, t-test, 2 sided

99. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): HDL-Z
Description: HDL-Z is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nm
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nm | 0.053 (0.060) | 0.089 (0.055)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.384, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.112, t-test, 2 sided

100. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): S-HDL-P
Description: S-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µmol/L | 0.434 (0.910) | 0.118 (0.902)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.636, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.896, t-test, 2 sided

101. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): M-HDL-P
Description: M-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µmol/L | 0.203 (0.793) | 0.500 (0.830)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.800, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.551, t-test, 2 sided

102. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): LM-HDL-P
Description: LM-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µmol/L | 0.595 (0.761) | 1.061 (0.757)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.440, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.170, t-test, 2 sided

103. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): L-HDL-P
Description: L-HDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µmol/L | 0.332 (0.301) | 0.503 (0.288)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.278, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.089, t-test, 2 sided

104. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): LDL-C
Description: LDL-C is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
mg/dL | 1.158 (4.414) | 4.737 (4.358)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.795, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.284, t-test, 2 sided

105. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): LDL-P
Description: LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | 5.605 (36.791) | 78.105 (34.245)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.880, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.028, t-test, 2 sided

106. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): LDL-Z
Description: LDL-Z is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nm
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nm | 0.037 (0.113) | -0.118 (0.091)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.746, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.199, t-test, 2 sided

107. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): S-LDL-P
Description: S-LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | -9.184 (38.768) | 53.605 (24.610)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.814, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.036, t-test, 2 sided

108. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): L-LDL-P
Description: L-LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µmol/L | 25.105 (36.371) | -1.658 (32.843)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.494, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.960, t-test, 2 sided

109. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): VL-LDL-P
Description: VL-LDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | 9.605 (33.684) | 71.605 (31.228)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.777, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.028, t-test, 2 sided

110. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): VLDL-P
Description: VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | 4.934 (4.144) | 0.645 (3.879)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.241, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.869, t-test, 2 sided

111. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): VLDL-Z
Description: VLDL-Z is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nm
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nm | -0.039 (1.347) | 3.113 (1.177)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.977, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.012, t-test, 2 sided

112. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): VLDL-TG
Description: VLDL-TG is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
mg/dL | 3.553 (6.558) | 10.458 (5.958)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.591, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.088, t-test, 2 sided

113. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): S-VLDL-P
Description: S-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | 2.913 (2.548) | -1.842 (2.876)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.260, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.526, t-test, 2 sided

114. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): M-VLDL-P
Description: M-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | 1.753 (2.866) | 1.008 (2.507)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.545, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.690, t-test, 2 sided

115. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): LM-VLDL-P
Description: LM-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | 1.676 (2.725) | 2.432 (2.534)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.542, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.344, t-test, 2 sided

116. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): L-VLDL-P
Description: L-VLDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | 0.095 (0.912) | 1.724 (0.787)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.918, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.035, t-test, 2 sided

117. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): IDL-P
Description: IDL-P is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
nmol/L | -12.316 (18.508) | 18.211 (27.738)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.510, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.516, t-test, 2 sided

118. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): ApoA1
Description: ApoA1 is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
mg/dL | 5.792 (2.799) | 5.272 (3.011)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.046, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.088, t-test, 2 sided

119. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): ApoB
Description: ApoB is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
mg/dL | 2.225 (2.568) | 3.360 (2.443)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.392, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.177, t-test, 2 sided

120. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): TRLTG
Description: TRLTG is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
mg/dL | 4.520 (8.180) | 14.465 (7.589)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.584, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.065, t-test, 2 sided

121. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): TRLC
Description: TRLC is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
mg/dL | 1.547 (1.902) | 2.598 (1.742)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.421, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.145, t-test, 2 sided

122. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): TRLP
Description: TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
nmol/L | 5.539 (10.787) | 8.555 (8.946)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.611, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.345, t-test, 2 sided

123. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): VS-TRLP
Description: VS-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
nmol/L | 0.619 (11.281) | 7.361 (9.130)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.957, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.425, t-test, 2 sided

124. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): S-TRLP
Description: S-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
nmol/L | 2.714 (6.936) | -2.990 (7.959)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.698, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.709, t-test, 2 sided

125. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): M-TRLP
Description: M-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
nmol/L | 1.976 (2.141) | 2.204 (1.768)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.362, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.221, t-test, 2 sided

126. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): L-TRLP
Description: L-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
nmol/L | 0.233 (0.976) | 1.981 (0.960)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.813, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.046, t-test, 2 sided

127. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): VL-TRLP
Description: VL-TRLP is a marker of lipid function and metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
nmol/L | -0.003 (0.011) | -0.002 (0.008)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.752, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.808, t-test, 2 sided

128. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Insulin
Description: Insulin is a marker of glucose metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
ng/ml | 421.436 (361.693) | 330.523 (334.064)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.251, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.329, t-test, 2 sided

129. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): HOMA-IR
Description: as for outcome 53
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: index
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
index | 1.814 (1.438) | 0.753 (1.471)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.215, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.612, t-test, 2 sided

130. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Glucose
Description: Glucose is a marker of glucose metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
mg/dL | 8.032 (7.746) | 2.604 (6.386)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.307, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.686, t-test, 2 sided

131. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): DRI
Description: as for outcome 55
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: index
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
index | -2.834 (1.875) | 1.765 (1.865)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.139, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.350, t-test, 2 sided

132. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): LP-IR
Description: as for outcome 56
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: index
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
index | -1.158 (3.219) | 2.684 (2.474)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.721, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.285, t-test, 2 sided

133. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Leptin
Description: Leptin is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
ng/ml | -498.841 (1993.620) | 304.320 (1149.111)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.804, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.793, t-test, 2 sided

134. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Adiponectin
Description: Adiponectin is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 38 | 38
µg/ml | -2.106 (1.975) | 1.268 (1.353)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.293, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.355, t-test, 2 sided

135. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Fetuin A
Description: Fetuin A is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µg/ml
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µg/ml | -53.518 (31.837) | 36.686 (26.223)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.101, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.170, t-test, 2 sided

136. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Citrate
Description: Citrate is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -5.547 (3.643) | -4.766 (3.684)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.137, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.204, t-test, 2 sided

137. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Valine
Description: Valine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -12.589 (7.799) | 6.269 (7.017)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.115, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.378, t-test, 2 sided

138. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Leucine
Description: Leucine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -8.223 (5.198) | 1.313 (5.585)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.122, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.815, t-test, 2 sided

139. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Isoleucine
Description: Isoleucine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -3.541 (3.519) | 5.203 (4.025)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.321, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.204, t-test, 2 sided

140. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Alanine
Description: Alanine is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | 23.209 (24.631) | 39.496 (28.893)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.352, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.180, t-test, 2 sided

141. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): BCAA
Description: BCAA is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -24.353 (14.136) | 12.785 (14.474)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.094, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.383, t-test, 2 sided

142. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Ketone Bodies
Description: Ketone Bodies are markers of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -79.323 (33.786) | -48.175 (42.608)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.024, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.266, t-test, 2 sided

143. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Beta Hydroxybutyrate
Description: Beta Hydroxybutyrate is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -48.450 (22.919) | -38.228 (29.792)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.042, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.208, t-test, 2 sided

144. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Acetoacetic Acid
Description: Acetoacetic Acid is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | 1.616 (2.094) | 0.993 (1.936)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.446, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.611, t-test, 2 sided

145. Secondary Outcome: Changes in Cardiometabolic Markers Between Week 52 and Earlier Time Points (Baseline and Week 16): Acetone
Description: Acetone is a marker of adipose dysfunction and general metabolism.
Time Frame: After the completion of week 52 visit by all study participants.
Population: The number of subjects analyzed reflect availability of analyzable samples.
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Week 52 vs. Baseline | Week 52 vs. Week 16
Number analyzed (Participants) | 37 | 37
µmol/L | -32.489 (12.565) | -10.939 (12.987)
Statistical Analysis 1: Comparison: Week 52 vs. Baseline; Test type: Superiority; p = 0.014, t-test, 2 sided
Statistical Analysis 2: Comparison: Week 52 vs. Week 16; Test type: Superiority; p = 0.405, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to Week 52
Arm/Group | Apremilast
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 6/70
Other Adverse Events (participants affected / at risk) | 31/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=70)
Stroke (Vascular disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Soft tissue mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Mildly FDG avid amorphous soft tissue mass in the left breast
Hospitalization due to fall (General disorders) | 2 (2)
Fracture due to fall (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast (N=70)
Nausea (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 11
Headache (General disorders) | 11
Upper respiratory infection (Infections and infestations) | 5
Dizziness (General disorders) | 4

LIMITATIONS AND CAVEATS:
The lack of placebo control; The number of biomarkers assessed may result in alpha error given the large number of pathways interrogated and thus the cardiometabolic biomarkers may be considered exploratory; Only surrogate markers evaluated and not actual clinical events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03082729/Prot_SAP_000.pdf